CLINICAL TRIAL: NCT03514693
Title: A Multicenter, Randomized Controlled, Non-inferiority Trial Investigating Efficacy and Safety of Pulmonary Vein Isolation Alone for Recurrence Prevention Compared to Extensive Ablation in Patients With Persistent Atrial Fibrillation
Brief Title: Efficacy of Pulmonary Vein Isolation Alone in Patients With Persistent Atrial Fibrillation
Acronym: EARNEST-PVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Osaka Cardiovascular Conference (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14377-8
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation; Catheter Ablation; Recurrence
Keywords: Persistent atrial fibrillation; non-inferiority trial
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI alone (Active Comparator): PVI, and ablation for AF triggers from non-PV foci, the cavotricuspid isthmus, clinical coexisting tachyarrhythmia such as atrial flutter (AFL), atrial tachycardia (AT), and supraventricular tachycardia, if necessary
  Interventions: Procedure: PVI
- PVI plus additional ablation (Placebo Comparator): PVI, additional CFAE or linear ablation after PVI, and ablation for AF triggers from non-PV foci, the cavotricuspid isthmus, clinical coexisting tachyarrhythmia such as atrial flutter (AFL), atrial tachycardia (AT), and supraventricular tachycardia, if necessary
  Interventions: Procedure: PVI plus additional ablation

INTERVENTIONS:
Procedure: PVI — Ipsilateral circumferential PVI is the recommended PVI strategy. The success of PVI is defined as the achievement of the dissociation of PV potentials in all PVs. Disappearance of PV potentials is reconfirmed at the end of the procedure, a minimum of 20 minutes after the initial success of PVI.
  Arms: PVI alone
Procedure: PVI plus additional ablation — In addition to PVI, CFAE ablation, linear ablation, or both; the choice of which is decided by the physician
  Arms: PVI plus additional ablation

SUMMARY:
This study examines non-inferiority of pulmonary vein isolation (PVI) for persistent atrial fibrillation (AF) to extensive ablation; and reveals the effect of the presence or origin of AF trigger on outcomes of catheter ablation.

DETAILED DESCRIPTION:
Study design The EARNEST-PVI trial is a prospective, multicenter, randomized, open-label non-inferiority trial in which patients with persistent AF will undergo ablation. After providing written informed consent at each hospital, patients who are eligible for the trial will be randomized to either PVI alone or PVI plus additional ablation. Left atrial dimensions will be the only adjustment factor considered in dynamic allocation to avoid bias. Patients randomized to the PVI alone group will be treated with PVI, while patients randomized to the PVI plus additional ablation group will receive additional complex fractionated atrial electrogram or linear ablation after PVI. Ablation for AF triggers from non-PV foci, the cavotricuspid isthmus, clinical coexisting tachyarrhythmia such as atrial flutter (AFL), atrial tachycardia (AT), and supraventricular tachycardia will be allowed in both groups. Patients will be followed up 1, 3, 6, 9, and 12 months after the procedure. The primary endpoint of the study is the recurrence of AF documented by scheduled or symptom-driven ECG during 1 year after the procedure. "Recurrence of AF" is defined as the documentation of any atrial arrhythmia including AF, AFL, and/or AT lasting ≥ 30 seconds by ECG or other appropriate tests. The sample size and randomization are specified based on the concept of non-inferiority to achieve the primary objective. The recurrence rate of AF was assumed to be 40% in both groups and a non-inferiority margin of 10% was calculated by referring to the previous studies. Therefore, a sample size of 256 subjects in each group is required with a power of 80% and significance level of 5% considering some dropouts. The statistical evaluation will be carried out according to the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a first-time ablation procedure for persistent AF

Exclusion Criteria:

* Patients with long-standing persistent AF lasting ≥ 5 years
* Patients with left atrial dimension ≥ 50 mm by 2-dimensional echocardiography
* Patients with valvular AF (defined as the presence of mitral or aortic stenosis or regurgitation with a history of rheumatic fever or implantation of artificial heart valves)
* Patients who underwent prior cardiac surgery
* Patients receiving hemodialysis
* Patients with heart failure (left ventricular ejection fraction < 30% and NYHA class ≥ III)
* Patients receiving antiarrhythmic agents before the ablation procedure (within 60 days for amiodarone, or 5 half-lives for other drugs)
* Patients who are not considered to be suitable candidates by the attending physician

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
recurrence of AF documented by scheduled or symptom-driven ECG during 1 year after the procedure | 1 year
  "Recurrence of AF" is defined as the documentation of any atrial arrhythmia including AF, AFL, and/or AT lasting ≥ 30 seconds by ECG or other appropriate tests.

SECONDARY OUTCOMES:
cardiovascular events | 1 year
  death (and/or cause of death), or symptomatic cerebral infarction
The effect of the presence or absence of AF trigger foci | 1 year
  recurrence of AF according to the presence or absence of AF trigger foci

CONTACTS AND LOCATIONS:
Overall Officials: Yasushi Sakata, MD, PhD, Principal Investigator — Department of Cardiovascular Medicine, Osaka University Graduate School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okada M, Inoue K, Tanaka N, Masuda M, Watanabe T, Makino N, Egami Y, Oka T, Minamiguchi H, Miyoshi M, Kanda T, Matsuda Y, Kawasaki M, Tanaka K, Hirao Y, Hikoso S, Sunaga A, Dohi T, Nakatani D, Okada K, Sotomi Y, Sakata Y; Osaka Cardiovascular Conference (OCVC)-Arrhythmia Investigators*. Impact of Initial Extensive Ablation on Left Atrial Gaps During Redo Procedures and Subsequent Outcomes in Persistent Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2025 Jun;18(6):e013612. doi: 10.1161/CIRCEP.124.013612. Epub 2025 Jun 2. PMID 40455466
- [Derived] Matsuoka Y, Sotomi Y, Hikoso S, Sunaga A, Nakatani D, Okada K, Dohi T, Sato T, Kida H, Sakamoto D, Kitamura T, Tanaka N, Masuda M, Watanabe T, Minamiguchi H, Egami Y, Oka T, Miyoshi M, Okada M, Matsuda Y, Kawasaki M, Inoue K, Sakata Y; OCVC-Arrhythmia Investigators. Extensive ablation for elderly patients with persistent atrial fibrillation: insights from the EARNEST-PVI prospective randomized trial. J Cardiol. 2025 Apr;85(4):301-308. doi: 10.1016/j.jjcc.2024.09.001. Epub 2024 Sep 7. PMID 39251131
- [Derived] Matsunaga-Lee Y, Inoue K, Tanaka N, Masuda M, Watanabe T, Makino N, Egami Y, Oka T, Minamiguchi H, Miyoshi M, Okada M, Kanda T, Matsuda Y, Kawasaki M, Kawanami S, Sugae H, Ukita K, Kawamura A, Yasumoto K, Tsuda M, Okamoto N, Yano M, Nishino M, Sunaga A, Sotomi Y, Dohi T, Nakatani D, Hikoso S, Sakata Y; Osaka Cardiovascular Conference (OCVC) Arrhythmia Investigators. Appropriate Selection of Substrate Ablation for Persistent Atrial Fibrillation Using Intraprocedural Assessment. Circ J. 2024 Jun 25;88(7):1068-1077. doi: 10.1253/circj.CJ-23-0936. Epub 2024 May 30. PMID 38811199
- [Derived] Sato T, Sotomi Y, Hikoso S, Nakatani D, Mizuno H, Okada K, Dohi T, Kitamura T, Sunaga A, Kida H, Oeun B, Egami Y, Watanabe T, Minamiguchi H, Miyoshi M, Tanaka N, Oka T, Okada M, Kanda T, Matsuda Y, Kawasaki M, Masuda M, Inoue K, Sakata Y; Osaka Cardio Vascular Conference (OCVC)-Arrhythmia Investigators *. DR-FLASH Score Is Useful for Identifying Patients With Persistent Atrial Fibrillation Who Require Extensive Catheter Ablation Procedures. J Am Heart Assoc. 2022 Aug 16;11(16):e024916. doi: 10.1161/JAHA.121.024916. Epub 2022 Aug 5. PMID 35929474
- [Derived] Curran L, Nah G, Marcus GM, Tseng Z, Crawford MH, Parikh NI. Clinical Correlates and Outcomes of Methamphetamine-Associated Cardiovascular Diseases in Hospitalized Patients in California. J Am Heart Assoc. 2022 Aug 16;11(16):e023663. doi: 10.1161/JAHA.121.023663. Epub 2022 Aug 1. PMID 35912709
- [Derived] Inoue K, Hikoso S, Masuda M, Furukawa Y, Hirata A, Egami Y, Watanabe T, Minamiguchi H, Miyoshi M, Tanaka N, Oka T, Okada M, Kanda T, Matsuda Y, Kawasaki M, Hayashi K, Kitamura T, Dohi T, Sunaga A, Mizuno H, Nakatani D, Sakata Y; OCVC Arrhythmia Investigators. Pulmonary vein isolation alone vs. more extensive ablation with defragmentation and linear ablation of persistent atrial fibrillation: the EARNEST-PVI trial. Europace. 2021 Apr 6;23(4):565-574. doi: 10.1093/europace/euaa293. PMID 33200213
- See also: UMIN-CTR — https://upload.umin.ac.jp/cgi-open-bin/ctr_e/ctr_view.cgi?recptno=R000022454